CLINICAL TRIAL: NCT01422564
Title: A Randomized Multicentre Clinical Trial Comparing The Metal on Metal Hip System Versus The Metal on Highly Crossed Linked Polyethylene System
Brief Title: Metal on Metal Versus Metal on Highly Crossed Linked Polyethylene Sytem
Acronym: MOM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Components were recalled by Depuy
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RL 006
Record Dates: First submitted 2011-08-12; First posted 2011-08-24 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Congenital Dysplasia of the Hip; Ankylosing Spondylitis; Post-traumatic; Arthrosis; Injury of Hip and Thigh
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Hip Dislocation, Congenital; Spondylitis, Ankylosing; Hip Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metal on Metal (Active Comparator): Metal on Metal articulation system
  Interventions: Device: Metal on Metal Hip System
- HCLPC (Active Comparator): THA using Highly Cross Linked Polyethylene cup System
  Interventions: Device: Highly Cross Linked Polyethylene cup System

INTERVENTIONS:
Device: Metal on Metal Hip System — Total hip arthroplasty with a metal on metal component system
  Other Names: Depuy ASR
  Arms: Metal on Metal
Device: Highly Cross Linked Polyethylene cup System — Total hip arthroplasty with Highly Cross Linked Polyethylene cup System
  Other Names: Depuy Pinnacle Cup and Marathon liner
  Arms: HCLPC

SUMMARY:
This trial will evaluate the 36mm or greater metal head on metal hip system and compare it to the 32mm or 28mm metal head on polyethylene (liner) hip system in patients receiving a primary cementless total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects 65 years of age or older
* Subjects undergoing cementless hip arthroplasty. If a press fit metal articulation acetabulum is not possible; the modular cup system will be utilized with screw fixation and a metal head of the greatest diameter deemed appropriate and safe for the patient will be utilized.(At the discretion of the surgeon). The cup in this situation may have a metal or poly articulation. The patient will be followed as an intent to treat (the patient will be evaluated and included in the group as randomized)
* Subjects with, but not limited to, original diagnoses of osteoarthritis, avascular necrosis, rheumatoid arthritis, congenital dysplasia of the hip, ankylosing spondylitis, posttraumatic arthritis, and traumatic injury to the hip joint.
* Subjects who are able and willing to understand the conditions of informed consent, to participate in the study according to the protocol for the length of the expected term of follow-up, and to follow their physician's directions.

Exclusion Criteria:

* Subjects undergoing hip arthroplasty using a cemented femoral component and/or a bipolar prosthesis.
* Subjects with gross obesity, >45% over ideal body weight for age and height. Refer to Appendix A, Obesity Table.
* Subjects with active infections.
* Subjects with malignancy in the area of the involved hip joint.
* Subjects with a neuromuscular deficit that interferes with the subject's ability to limit weight bearing or places an extreme load on the implant during the healing period.
* Subjects with a diagnosis of Fibromyalgia
* Female subjects who are pregnant or may be pregnant.
* Subjects whom, as judged by the surgeon, are not capable of understanding the informed consent or the requirements of the protocol, or are reasonably unlikely to be compliant with the prescribed postoperative routine and the follow-up evaluation schedule.
* Subjects who have a known sensitivity to device materials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Revision Rate | 4 years

SECONDARY OUTCOMES:
Wear and osteolysis | 5-15 years
Harris Hip Score | immediate post-op, 6 months, 1 year, 2 years, 4 years
Dislocation Rate | 4 years
Complication Rate | 4 years
  All complications
Gait Analysis | 6 months and 1 year post-op
  Using the Walkabout portable gait monitor
Metal Ions | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, Principal Investigator — Nova Scotia Health Authority